CLINICAL TRIAL: NCT07203768
Title: Unmasking Polycythemia Vera in Long-Standing Essential Thrombocythemia: A ELN-Multicenter Study on Phenotypic Evolution and Clinical Outcomes
Brief Title: A ELN-Multicenter Study on Phenotypic Evolution and Clinical Outcomes
Acronym: ET2PV
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: ET2PV
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Polycythemia Vera; Thrombocythemia
MeSH Terms: conditions — Polycythemia Vera; Thrombocytosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ET to PV patients: Patients JAK2V617F positive and who have progressed to PV by 31/12/2020.
- ET patients: Patients JAK2V617F positive who did not progress to PV after a comparable period of time. This control group will be selected using a 1:1 matched case-control design.
- PV de novo patients: Patients diagnosed with de novo PV (no progression from previous ET). This control group will be recruited using a 1:1 matching procedure.

SUMMARY:
International multicenter retrospective observational study consisting of two parts: a nested case-control study (part A) and a comparative retrospective cohort study (part B).

DETAILED DESCRIPTION:
The study will include ET patients (diagnosed according to "International consensus classification of myeloid neoplasms and acute leukemias - 2022" criteria) who are JAK2V617F positive and have progressed to PV (diagnosed according to "International consensus classification of myeloid neoplasms and acute leukemias - 2022" criteria) by 31/12/2020. The date of PV diagnosis will be defined as the index date and this group of patients will be defined as ET-to-PV cases.

Part A - Nested case-control study Controls for ET-to-PV cases will be patients diagnosed with ET, according to the "International consensus classification of myeloid neoplasms and acute leukemias - 2022" criteria, JAK2V617F positive who did not progress to PV after a comparable period of time. This control group will be selected using a 1:1 matched case-control design.

For each patient who progressed to PV (case), a control will be selected with the following characteristics:

* year of ET diagnosis (+/-2 years as compared to the date of the case);
* age at ET diagnosis (+/-3 years as compared to the age of the case);
* duration of ET disease (+/-2 years as compared to the period between the diagnosis of ET and the index date of the respective case).

Part B - Comparative retrospective cohort study

Patients diagnosed with de novo PV (no progression from previous ET) according to the "International consensus classification of myeloid neoplasms and acute leukemias - 2022" data criteria, will be recruited using a 1:1 matching procedure according to the following characteristics:

* year of PV diagnosis (+/-2 years as compared to the date of the case);
* age at PV diagnosis (+/-3 years as compared to the age of the case);
* duration of PV disease (+/-2 years as compared to the period between PV diagnosis and the last follow-up of the respective case).

Furthermore, to have at least 5 years of follow-up, de novo PV patients must be diagnosed no later than 2020.

ELIGIBILITY:
Inclusion Criteria:

- ET patients (diagnosed according to "International consensus classification of myeloid neoplasms and acute leukemias - 2022" criteria) who are JAK2V617F positive and have progressed to PV (diagnosed according to "International consensus classification of myeloid neoplasms and acute leukemias - 2022" criteria) by 31/12/2020. The date of PV diagnosis will be defined as the index date and this group of patients will be defined as ET-to-PV cases.

Exclusion Criteria:

* None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nested case-control study: the prevalence of at least one of the following proliferative conditions in the control group, a neutrophil/lymphocyte ratio (N/L ratio) above the median, an LDH above the median, being JAK2V617F homozygous and having splenomegaly.
  Comparative retrospective cohort study: it is known that the incidence of the composite outcome (vascular events, cancers, progression to myelofibrosis, progression to acute myeloid leukemia, death) in PV de novo patients.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Nested case-control study | Up to the baseline
  To identify proliferative risk factors for progression from ET to PV in JAK2V617F positive patients.
Comparative retrospective cohort study | Up to the baseline
  To evaluate the different disease prognosis in ET patients who have progressed to PV compared to de novo PV patients.

SECONDARY OUTCOMES:
Nested case-control study | At the time of progression
  To describe characteristics of ET patients who progressed to PV, including the timing of progression.
Comparative retrospective cohort study | At the time of progression
  To compare the incidence of different outcomes (vascular events, progression to myelofibrosis, progression to acute myeloid leukaemia, tumours, death) in ET patients who progressed to PV and in de novo PV patients.

CONTACTS AND LOCATIONS:
Overall Officials: TIZIANO BARBUI, MD, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (25):
- Mayo Clinic, Rochester, Minnesota, United States
- Germany (3):
  - University Hospital Halle, Halle
  - Hannover Medical School, Hanover
  - University Clinic for Hematology, Oncology, Hemostaseology and Palliative Care Johannes Wesling Medical Center, Minden
- Italy (18):
  - Divisione Ematologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Divisione Ematologia, Ospedale San Bortolo, Vicenza, Veneto
  - A.S.O. SS. Antonio e Biagio e C.Arrigo, SC Ematologia, Alessandria
  - ASST Papa Giovanni XXIII, SC Ematologia, Bergamo
  - ASST-Spedali Civili, Brescia
  - Ospedale Businco, Cagliari
  - AOU Policlinico Vittorio Emanuele - PO Gaspare Rodolico, Catania
  - AOU Careggi, Divisione di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda, Divisione di Ematologia, Milan
  - Fondazione IRCCS Cà Grande - Op. Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - ASST MONZA Ospedale San Gerardo Clinica Ematologica, Monza
  - Azienda Ospedaliera Universitaria Federico II di Napoli Divisione di Ematologia e Trapianti del Midollo, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara SCDU Ematologia, Novara
  - Presidio Ospedaliero di Pescara, Pescara
  - Fondazione Policlinico Universitario Gemelli, Roma
  - Umberto I Policlinico, Roma
  - Azienda Ospedaliera Universitaria Integrata - Ospedale Borgo Roma, Unità di Ematologia, Verona
- Spain (2):
  - IDIBAPS, Hospital clinic, Barcelona
  - 12 Octubre University Hospital, Madrid
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom